CLINICAL TRIAL: NCT04104009
Title: The Relation Between Midwifery Education of Pregnant Women and Listening to Classical Music With the Mode of Delivery, the Length of Breastfeeding and the Incidence of Psychic Symptoms: RCT
Brief Title: The Relation Between Midwifery Education and Listening to Classical Music With the Mode of Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Mostar (Other)
Responsible Party: Principal Investigator, Roberta Perkovic, Head nurse of the department of women's diseases and childbirth, University of Mostar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMostar
Record Dates: First submitted 2019-09-19; First posted 2019-09-26 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Delivery Mode; Pain Score; Breastfeeding Rate; Mental Health Issue; Apgar Score
Keywords: midwifery; education; pregnancy; delivery mode; music therapy; breastfeeding; pain score; postnatal mental health; Apgar score
MeSH Terms: conditions — Breast Feeding | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The sample is suitable, pregnant women in the second and third trimester of pregnancy who will give birth in a maternity ward County Hospital "Dr. Mihovil Sucic" Livno from February 2019 to the beginning of September 2019.
  By randomization, the respondents will be divided into two groups:
  1. Interventional group- a group where group education, breathing exercise and listening to classical music will be conducted.
  2. Control group - a group who will spend the pregnancy without education, listening to classical music and breathing exercises.
  Both groups are subject to inclusion and exclusion criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): In the exam group there will be group training for four meetings of one hour each.
  After completing the training program with the test group, a break of 5 weeks will follow, during which a new test and control group will be formed. The procedure will be carried out until the estimated sample size (99 subjects per group) is met.
  Interventions: Other: Education
- Control group (Active Comparator): In the control group there will not be any group training.
  Interventions: Other: No education

INTERVENTIONS:
Other: Education — Following the randomization process, group education of pregnant women will be conducted through four one-hour meetings.
  Education program: teaching about the basics of childbirth physiology, visit to the maternity ward with the aim of reducing the fear of childbirth, applying the deep inhale and exhale exercise in the first birth stage, applying the classical music listening technique that will continue until the end of pregnancy daily (in the evenings before bedtime) (for 15 minutes), teaching and applying techniques for successful breastfeeding, maternal and infant health care after delivery. The training program will be implemented so that after 4 workshops a 5-week break will be taken. At the end of the program, the educator arranges with the respondents a weekly telephone check (for the sake of communication quality) to inform them of adherence to the agreed classical music listening.Pregnant women who do not meet expectations will be excluded from the study.
  Arms: Interventional group
Other: No education — In the control group there will be no education, no breathing exercises and no listening to classical music.
  Arms: Control group

SUMMARY:
The emotional and psychological well-being of women influence the perception and experience of pregnancy and childbirth. Pregnant women with a fear of childbirth are more likely to give birth by caesarean section. An increased risk of obstetric interventions such as planned and emergency caesarean section has been determined. Childbirth education is an intervention that has a major impact on maternity outcomes and birth experience

DETAILED DESCRIPTION:
The emotional and psychological well-being of women significantly affects the perception and experience of pregnancy and childbirth. Pregnant women with a fear of childbirth are more likely to give birth by caesarean section. An increased risk of obstetric interventions such as planned and emergency caesarean section was also identified. Childbirth education is an intervention that has a great impact on birth outcomes and childbirth experiences.

A Cochrane systematic review found that the effects of antenatal education on childbirth and parenting are quite unknown. In a longitudinal cohort study, on a sample of 576 women, Bossano et al. investigated the impact of the vaginal birth method and the experience experienced on health after a decade. It was found that women with caesarean section were significantly more distressed than those who had delivered vaginally, and that the experience of childbirth remains in the memory even after a decade.

A randomized controlled study conducted in Australia by Fenwick et al. divided a sample of 339 pregnant women into a test and control group measured the impact of midwifery education on outcomes in childbirth, breastfeeding and the development of postpartum depression. Pregnant women of the interventional group received individual psychoeducation training by midwives in the second trimester of pregnancy. The control group did not undergo individual training. Finally, 184 female respondents with duly completed questionnaires were included in the analysis. In comparison with the control group, the caesarean section rate in the interventional was clinically but not statistically significantly lower (by 8%), and the need for an emergency caesarean section in the test group was less than 7%. There was no difference in the assessment of postpartum depression between the two groups. At 6 weeks postpartum, there was no statistically significant difference in the infant's diet between the two groups. In the interventional group, 83.5% were breastfed and 78.5% in the control group. It was concluded that the psychoeducation of pregnant women had the effect of reducing the overall rate of caesarean section. The impact of education on psychosocial health was found in a randomized controlled study called "Mindfulness - based program on the psychological health of pregnant women" in a sample of 104 women, divided into an interventional and control group. Pregnant women in the interventional group attended an eight-week program in groups between 13 and 26 weeks of gestation and used audio recordings at home, and had statistically significantly lower levels of stress and depression compared to the control group when measured at 36 weeks of gestation.

The use of deep inhalation and exhalation breathing exercises has proven effective in reducing the perception of pain in childbirth. A randomized clinical trial by Yuksel et al. in a sample of 250 pregnant women divided into test and control groups, the aim was to determine the effectiveness of the exercise on the perception of pain and the impact on the Apgar score of the infant after 1 minute. Pregnant women underwent a series of exercise training sessions and practiced during the first delivery phase to reduce stress and relaxation. There was a statistically significant difference in the lower perception of pain in the interventional group compared to the control group. A VAS scale of pain was used to assess pain. There was no statistically significant difference in the value of the Apgar score.

The therapeutic effects of listening to music on maternal and infant health have been proven in numerous studies. A lower incidence of anxiety and depression in women, a lower perception of pain during childbirth, a higher oxygen saturation in a newborn infant, and longer breastfeeding were found. A unique package with selected music has not been defined, but the choice is left to the creativity and knowledge of health professionals. A statistically significantly lower level of pain and anxiety at all measured time intervals was determined by a study in which a test group of 80 first-timers listened to music of their choice during childbirth compared to a control group who underwent childbirth without listening to music.

Based on the results of various studies, it can be concluded that the influence of antenatal education on the reduction of the rate of caesarean section in relation to vaginal delivery and the perception of pain during childbirth. Listening to classical music and breathing exercises significantly contribute to the reduction of labor pain, affecting the length of breastfeeding and the mental health of women in the maternity ward. An area requiring research is the fear of childbirth and its consequent impact on both maternity outcomes and the mental health of women in the ward.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Territory of Herceg-Bosna County
* Monitoring pregnancy in the competent Health Centers and private gynecological surgeries

Exclusion Criteria:

* Minor pregnant women
* Pregnant women in the first trimester of pregnancy
* Pregnant women after the 34th week of gestation
* Multiple pregnancies
* Pregnant women having a cesarean delivery in their anamnesis
* Pregnant women with psychiatric diagnosis
* Pregnancies at-risk
* Incomplete or illegally filled questionnaires
* Pregnant women who did not listen to classical music the agreed way
* Delivery of a stillborn baby

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 198 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Delivery Mode | up to 10 months
  caesarean section or vaginal birth

SECONDARY OUTCOMES:
Apgar score | up to 10 months
  The Apgar score is a test given to newborns soon after birth. In the test, five things are used to check a baby's health. Each is scored on a scale of 0 to 2, with 2 being the best score:
  1. Appearance (skin color)
  2. Pulse (heart rate)
  3. Grimace response (reflexes)
  4. Activity (muscle tone)
  5. Respiration (breathing rate and effort) Scores are between 10 and 0. The test is given in the first and fifth minute. A baby who scores a 7 or above on the test is considered in good health. Perfectly healthy babies sometimes have a lower-than-usual score, especially in the first few minutes after birth.
  Scores of 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts.
Pain score | up to 10 months
  A Visual Analogue Scale (VAS) is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.
  The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations. Recall period for items varies, but most commonly respondents are asked to report "current" pain intensity or pain intensity "in the last 24 hours.
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post- surgical patients have been recommended: no pain (0-0,4 cm), mild pain(0,5-4,4 cm), moderate pain (4,5-7,4 cm), and severe pain (7,5-10 cm).
Breastfeeding | up to 10 months
  Establishment of breastfeeding 6 weeks after maternity discharge. It is measured by a self-administered breastfeeding questionnaire. The questionnaire was created for research purposes. It contains 5 questions. The questionnaire has been sent to the patients six weeks after delivery. The purpose of the questionnaire is to claim answers about modes of feeding of newborns after six weeks (exclusive/not exclusive breastfeeding), to find out about support of women after delivery, to find reason of giving up on exclusive breastfeeding (if they gave up), to determine who had the gratest influence in their attitude about breastfeeding.
Psychic symptoms | up to 10 months
  The Symptom Checklist-90-R (SCL-90-R) is a relatively brief self-report psychometric instrument (questionnaire) published by the Clinical Assessment division of the Pearson Assessment & Information group. It is designed to evaluate a broad range of psychological problems and symptoms of psychopathology. It consists of 90 items and takes 12-15 minutes to administer, yielding nine scores along primary symptom dimensions and three scores among global distress indices. The primary symptom dimensions that are assessed are somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, and a category of "additional items" which helps clinicians assess other aspect of the clients symptoms (e.g. item 19, "poor appetite"). The three indices are global wellness index, hardiness, and symptom free. It is one of the most widely used measures of psychological distress in clinical practice and research.

CONTACTS AND LOCATIONS:
Locations (1):
- County Hospital 'Dr. fra Mihovil Sucic', Livno, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No